CLINICAL TRIAL: NCT02042924
Title: Pilot Study of Multi-Modality Imaging in Patients With Hematologic Malignancies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Updating protocol and consents
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013NTLS100; MT2013-28R (Other: University of Minnesota Blood and Marrow Transplant Program)
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Hematologic Malignancy
Keywords: Leukemia; Lymphoma; Myeloma; Myelodysplastic Syndrome
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imaging studies (Experimental): Subjects will have a FLT PET/CT and a MRI prior to starting the preparative regimen for transplant and another of each scan 100 days after transplant.
  Interventions: Radiation: FLT PET/CT; Device: MRI

INTERVENTIONS:
Radiation: FLT PET/CT — Functional marrow imaging using the FLT PET/CT will be performed prior to preparative for HSCT and approximately 3 months post-transplant (Day 100 +/- 5 days).
Device: MRI — MRI imaging will be performed prior to preparative for HSCT and approximately 3 months post-transplant (Day 100 +/- 5 days).

SUMMARY:
This is a pilot sub-study of patients receiving myeloablative transplant using total body irradiation (TBI) or total marrow irradiation (TMI) in their preparative regimen. The objective of this stub-study is to estimate the heterogeneity in cellular proliferation (FLT-PET uptake) as well the heterogeneity in marrow composition distribution (measured using whole body water-fat MRI) using positron emission tomography imaging. This will be used to design future trials as well as to determine the feasibility of PET and MRI imaging.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hematologic malignancy and fitting into one of the following categories:

  * Newly diagnosed and/or day 14 post-induction chemotherapy
  * Relapsed, including relapse after hematopoietic cell transplant
  * Planned hematopoietic cell transplant (if enrolling at "close") or within 100 days post hematopoietic cell transplant (if enrolling post-transplant) with a preparative regimen that includes either total marrow irradiation (TMI) or total body irradiation (TBI)
  * Undergoing natural killer cell therapies (with or without subsequent transplant)
* Aged 18 years and older
* Not pregnant - women of childbearing potential will have a confirmatory pregnancy test prior to each imaging per routine procedures
* Adequate renal function (estimated glomerular filtration rate > 60 ml/min) as determined by a serum creatinine level performed as a part of standard of care within 7 days of imaging
* Able and willing to provide written consent

Exclusion Criteria:

* Otherwise eligible patients meeting one or more of the contraindicates for an MRI, may enroll in the study without undergoing the MRI:

  * ferromagnetic implants
  * history of shrapnel or shot gun injury
  * too large to fit in the magnet (approximate body mass index ≥ 40)
  * cardiac pacemakers or other implanted devices that are not MR-compatible
  * claustrophobia
  * large tattoos

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanta K Hui, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imaging Studies
Started | 2
Completed | 1
Not Completed | 1
Not completed — Early Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Imaging Studies
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Difference in Percentage of Proliferating Bone Marrow Between Baseline and 100 Days
Description: The difference in percentage of proliferating bone marrow will be calculated for the following sites: skull, proximal humeri, ribs, clavicles, cervical spine, thoracic spine, lumbar spine, sacrum, pelvis and proximal femur.
Time Frame: 100 days
Population: Only one patient was enrolled in each cohort and therefore any analysis would not be meaningful.
Arm/Group | Imaging Studies
Number analyzed (Participants) | 0

2. Primary Outcome: Difference in Water Fat
Description: The difference in the water-fat MRI between baseline and day 100 post transplant in L4 and femoral neck.
Time Frame: 100 days
Population: Only one patient was enrolled in each cohort and therefore any analysis would not be meaningful.
Arm/Group | Imaging Studies
Number analyzed (Participants) | 0

3. Primary Outcome: Percentage of Proliferating Bone Marrow in the Femur
Description: The difference in the percentage of proliferating bone marrow between baseline and day 100 post transplant in the femur
Time Frame: 100 days
Population: Only one patient was enrolled in each cohort and therefore any analysis would not be meaningful.
Arm/Group | Imaging Studies
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Imaging Studies
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imaging Studies (N=2)
Sweating (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No